CLINICAL TRIAL: NCT03348436
Title: Study on Left Atrial Function of Paroxysmal Supraventricular Tachycardia After Radiofrequency Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruiqin xie (Other)
Responsible Party: Sponsor-Investigator, Ruiqin xie, director of cardiology department, The Second Hospital of Hebei Medical University
Organization: The Second Hospital of Hebei Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: xierqdoctorSVT
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Paroxysmal Supraventricular Tachycardia
Keywords: paroxysmal supraventricular tachycardia; Left Atrial Function
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: A total of 100 patients with persistent，in whom successful RF ablation of slow pathway or accessory pathway was performed. Patients with atrial fibrillation, structural heart disease, ventricular arrhythmias, impaired left ventricular systolic function or on antiarrhythmics were excluded. All the patients had echocardiographic study before ablation 、1 day and 1 months after ablation.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with atrioventricular nodal reentrant tachycardia (Experimental): radiofrequency catheter ablation therapy
  Interventions: Procedure: radiofrequency ablation
- patients with atrioventricular tachycardia (Experimental): radiofrequency catheter ablation therapy
  Interventions: Procedure: radiofrequency ablation

INTERVENTIONS:
Procedure: radiofrequency ablation

SUMMARY:
This study to investigate the effects of RF ablation on left atrial systolic function in patients with atrioventricular nodal reentrant tachycardia (AVNRT) and atrioventricular tachycardia (AVRT).

DETAILED DESCRIPTION:
A total of 100 patients with persistent，in whom successful RF ablation of slow pathway or accessory pathway was performed. Patients with atrial fibrillation, structural heart disease, ventricular arrhythmias, impaired left ventricular systolic function or on antiarrhythmics were excluded. All the patients had echocardiographic study before ablation 、1 day and 1 months after ablation. Left atrial systolic function was assessed using atrial ejection force (AEF) according to Manning's formula (AEF = 0.5 x ρ x MA x A(2), r: blood density = 1.06 g/cm(3), MA: mitral orifice area [cm(2)], A: A wave velocity). The following left atrial dimensions were assessed: antero-posterior (LA-AP), infero-superior (LA-IS, long axis), medio-lateral (LA-ML, short axis). The correlations between AEF and electrophysiological parameters were analysed (VA - ventriculo-atrial conduction, VA/CL - tachycardia cycle length).

ELIGIBILITY:
Inclusion Criteria:

Patients with paroxysmal supraventricular tachycardia,includes atrioventricular reentrant tachycardia and atrioventricular nodal reentrant tachycardia， Age is >14 years

Exclusion Criteria:

Atrial fibrillation, Atrial tachycardia， Structural heart disease, Ventricular arrhythmias, Patients with impaired left ventricular systolic function or on antiarrhythmics

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Left Atrial Function of postoperative radiofrequency ablation. | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China